CLINICAL TRIAL: NCT03592212
Title: Phosphodiesterase 4 Gene Variant and Salbutamol Response in Persistent Childhood Asthma
Acronym: PEGASE2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16014
Record Dates: First submitted 2018-05-09; First posted 2018-07-19 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Asthma
Keywords: Asthma; Salbutamol response; Phosphodiesterase 4 variant; lung function; airflow limitation
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Saliva from patients will be collected using Oragen®. DNA OG-575 kit, (DNA Genotek, Kanata, Canada) and stored at room temperature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Salbutamol — Measurement of bronchodilator response (BDR)

SUMMARY:
This study is designed to investigate whether the Phosphodiesterase 4 gene variability could be implicated in the salbutamol responsiveness in asthmatic children.

DETAILED DESCRIPTION:
Patients from 6 to 18 years old with asthma and receiving a treatment by salbutamol according to the usual care will be recruited. Saliva from patients will be collected using Oragen®.DNA OG-575 kit.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-18 years
* Asthma: confirmed asthma symptoms (wheeze, cough, dyspnea, chest tightness) and evidence for variable airflow limitation (≥ 12% increase in post bronchodilator FEV1, or ≥ 20% decrease in FEV1 post methacholine)
* Spirometry prescribed for follow-up
* Airflow limitation: FEV1<80% and/or FEV1/FVC <80 pre-bronchodilator

Exclusion Criteria:

* no exclusion criteria

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 6-18 years old asthmatic patients consulting in the Department of Pediatric Pulmonology and Allergy of Necker University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
pre- and post-bronchodilator VEMS value | Day 0
  comparison of acute response to salbutamol calculated as the percentage difference between the pre- and post-bronchodilator VEMS value (BDR = 100 x [post-VEMS - pre-VEMS]/pre-VEMS) according to the genotype of the rs1504982

SECONDARY OUTCOMES:
Locating other regions of the PDE4 gene that may be associated with the response to salbutamol by gene mapping (using SNP tags) | Day 0
  To identify other SNPs on PDE4 associated with the response (BDR) to salbutamol in childhood asthma.
Screening other SNPs (other genes than PDE4) associated with the response to salbutamol in childhood asthma using SNP tags | Day 0
  To identify other genes that could be associated with the phenotype of interest (BDR) by tagging other genes.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEZMI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker -Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No